CLINICAL TRIAL: NCT01427465
Title: Brief Integrative Alcohol Interventions for Adolescents
Acronym: Brief
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left University of Florida
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: #2007-U-0085; R01AA009283 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2011-09-01 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Alcohol Abuse; Drug Abuse
Keywords: Brief; Image; Intervention; Adolescents; School
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Consult (Experimental): Consult
  Interventions: Behavioral: Brief Prevention Program Using Positive Image
- Newsletter (Experimental): Newsletter
  Interventions: Behavioral: Brief Prevention Program Using Positive Image
- Parent Letter (Experimental): Parent Letter
  Interventions: Behavioral: Brief Prevention Program Using Positive Image
- Control (Active Comparator): Control
  Interventions: Behavioral: Brief Prevention Program Using Positive Image

INTERVENTIONS:
Behavioral: Brief Prevention Program Using Positive Image — Consult
  Other Names: Consult
  Arms: Consult
Behavioral: Brief Prevention Program Using Positive Image — Control - Standard of Care
  Other Names: Control
  Arms: Control
Behavioral: Brief Prevention Program Using Positive Image — Newsletter
  Other Names: Newsletter
  Arms: Newsletter
Behavioral: Brief Prevention Program Using Positive Image — Parent Letter
  Other Names: Parent Letter
  Arms: Parent Letter

SUMMARY:
The primary aim of this research is to test the efficacy of innovative, brief alcohol abuse prevention strategies that integrate positive youth development messages and health risk messages for adolescents in high school settings. A secondary aim is to examine these strategies in various combinations as interventions and re-interventions (i.e., boosters) for sustaining or enhancing behavior change over time. These strategies are founded upon an emerging conceptual framework titled the Behavior-Image Model emanating from findings of our recent trials examining multiple behavior health interventions. The long-term objective of this project is to reduce alcohol abuse and problems among older high-risk adolescents for whom alcohol and drug use disparities exist, yet who are often overlooked in prevention research and services.

DETAILED DESCRIPTION:
A total of 921 adolescents from two diverse high schools in northeast Florida were randomized to receive either the: 1) in-person consult, 2) parent-youth letter, 3) adolescent newsletter, or 4) standard care control . Three-month, one-year and 18-month follow-ups are planned, with interventions to be implemented in rotating fashion as re-interventions immediately after three-month and one-year data collections. Plans for following year include the following: 1) collecting and analyzing 3-month post-intervention data to determine the effects of the initial consult, parent-youth and adolescent print strategies, intervention costs, and assess possible mediators and moderators of outcomes; 2) implementing the first round of re-interventions; 3) collecting and analyzing one-year post-baseline effects of re-interventions, determining costs and cost-effectiveness of the interventions/re-interventions, and assessing possible mediators and moderators of outcomes; and 4) implementing the second round of re-interventions.

ELIGIBILITY:
Inclusion Criteria:

* Can read English
* 10th and 11th grade high school students at participating sites

Exclusion Criteria:

* Cannot read English
* Not in 10th and 11th grade high school students at participating sites

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in alcohol, cigarette and marijuana use consumption from baseline to 3 months follow up. | Baseline to 3 months follow up
Change in alcohol, cigarette and marijuana use consumption from baseline to 12 months follow up. | Baseline to 12 months follow up
Change in alcohol, cigarette and marijuana use consumption from baseline to 18 months follow up. | Baseline to 18 months follow up

SECONDARY OUTCOMES:
Change in frequency of health promoting behaviors from baseline to 3 months follow up. | Baseline to 3 months follow up
Change in frequency of health promoting behaviors from baseline to 12 months follow up. | Baseline to 12 months follow up
Change in frequency of health promoting behaviors from baseline to 18 months follow up. | Baseline to 18 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Chudley E Werch, PhD, Principal Investigator — Addictive & Health Behaviors Research Institute, University of Florida
Locations (1):
- Addictive & Health Behaviors Research Institute, University of Florida, Jacksonville, Florida, United States